CLINICAL TRIAL: NCT07080281
Title: Evaluation of the Effectiveness of Virtual Reality Application During Cesarean Delivery in Pregnant Women Undergoing Spinal Anesthesia
Brief Title: Evaluating the Effectiveness of Virtual Reality Application in Caesarean Section
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Fatma Çelik, Nurse, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FC-AYBU-09-451
Record Dates: First submitted 2025-05-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Virtual Reality Pain Distraction; Birth Satisfaction; Vital Signs; Anxiety; Apgar Score; Virtual Reality
Keywords: labor pain; cesarean section; birth satisfaction; birth anxiety; apgar scores; virtual reality; hemodynamic parameters
MeSH Terms: conditions — Anxiety Disorders; Labor Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality group (Active Comparator): group using virtual reality glasses
  Interventions: Device: Oculus Meta Quest 2 All In-One model virtual reality glasses
- control group (No Intervention): group without virtual reality glasses

INTERVENTIONS:
Device: Oculus Meta Quest 2 All In-One model virtual reality glasses — During the caesarean section, Meta Quest 2 All In-One model virtual reality glasses from Oculus were used for 15 minutes. In this virtual environment, the licensed product video "Breathe- Relax and Meditate" was watched via the "Meta Horizon" application.
  Arms: virtual reality group

SUMMARY:
The aim of this study was to evaluate the effects of virtual reality intervention during cesarean delivery under spinal anesthesia on labor pain, anxiety, satisfaction and hemodynamic parameters in primiparous pregnant women.

The main questions it aims to answer are:

1. Is there a significant difference between the mean intraoperative pain scores of the pregnant women in the intervention group and those in the control group?
2. Is there a significant difference between the mean intraoperative anxiety scores of the pregnant women in the intervention group and those in the control group?
3. Is there a significant difference between the mean birth satisfaction scores of the pregnant women in the intervention group and those in the control group?
4. Is there a significant difference between the vital signs of pregnant women in the intervention group and those in the control group?
5. Is there a significant difference between the mean apgar scores of the pregnant women in the intervention group and those in the control group?

DETAILED DESCRIPTION:
The study was conducted in the cesarean section unit of a university hospital. Pregnant women who were planned for cesarean section and applied to the outpatient clinic for routine examinations such as non-stress test (NST) and monitoring of vital signs, ultrasound, laboratory tests, information about preoperative preparation (stopping oral intake 6-8 hours before cesarean section, antibiotic prophylaxis, not wearing jewelry, hair clips, contact lenses, artificial nails, nail polish, etc., and 48 hours of hospital stay in the postpartum period) were informed about the study and the "Research Inclusion Criteria Form" was applied. In order to assign equally to the intervention and control groups of pregnant women who met the inclusion criteria and volunteered, they were assigned numbers according to the order of their application to the outpatient clinic and simple random sampling method was used on the website https://randomizer.org/randomize. All pregnant women were informed about the purpose, content and duration of the study and their written consent was obtained. During the process in which the effectiveness of spinal anesthesia was evaluated, virtual reality glasses were applied to pregnant women in the intervention group for approximately 5 minutes and then removed to rest. The resting period lasted an average of 10 minutes, although it varied depending on the patient in whom the effect of spinal anesthesia was complete. The second application of the virtual reality glasses was applied for approximately 10 minutes from the opening of the surgical incision line until the head/extremity/rectum of the fetus was visible. The virtual reality glasses application was terminated at the moment the newborn was born. No intervention was made to the control group during these procedures. The virtual reality glasses applied to the intervention group during the cesarean delivery are the Meta Quest 2 All In-One model from the Oculus brand, which can be worn on the head. Thanks to its head-mountable feature, the glasses isolate the real world. Each of the glasses' lenses has a resolution of 1832x1920 pixels and a 360˚ field of view. The glasses are used by pairing them with the ''Meta Horizon'' application purchased from application markets. The "Breathe- Relax & Meditate" licensed product video, which can be purchased from the "Meta Horizon" application, will be played on the virtual reality glasses. This product includes videos with images of lakes, forests, waterfalls, beaches, and rivers, along with a meditation music background.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age and older,
* Turkish speaking,
* At least primary school graduate,
* Between 37th and 42nd weeks of pregnancy, primiparous and with a single fetus,
* No diagnosed psychiatric problem (anxiety disorder, bipolar disorder, schizophrenia, etc.),
* No epilepsy diagnosis,
* No hearing, vision or communication impairment,
* Spinal anesthesia planned,
* Pregnant women who volunteered to participate in the study were included.

Exclusion Criteria:

* Incomplete data collection forms,
* Participant's refusal to participate in the study at any stage,
* Use of general anesthesia/sedation during the cesarean section process,
* Only for pregnant women in the intervention group; not fully participating in the virtual reality glasses training, not using the virtual reality glasses for the desired duration, or having side effects of the virtual reality glasses (dizziness, headache, sweating, nausea, vomiting or eye strain) are the exclusion criteria from the study.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 55 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | Birth anxiety was assessed at two different times. The first; 6-12 hours before cesarean delivery, and the second; was during the cesarean section, between 6-15th minutes.
  Pregnancy, birth and the transition to parenthood are important milestones in a woman's life, both physically, emotionally and socially. A cesarean section is an anxious process because it is both a birth and a surgical intervention. Especially for those who are giving birth for the first time, fears that the mother will experience pain during birth and possible risks to the health of the mother and newborn increase the anxiety and concerns about this process. In the management of anxiety during pregnancy, birth and postpartum periods, pharmacological interventions are avoided due to their possible negative effects on the fetus. This situation increases the importance of using nonpharmacological methods in the management of anxiety. The minimum score obtained from the scale is 20, the maximum score is 80. A high score obtained from the scale means that anxiety is high. The cut-off score of the scale is 39-40.
Maternal Satisfaction Evaluation Scale (Cesarean Section) | Between 0-25th minutes of cesarean delivery
  It is reported that birth satisfaction is an important parameter in protecting mother-baby health. Therefore, birth satisfaction is one of the important indicators of the quality of health care provided. The World Health Organization recommends that a birth care should be organized and provided in order to ensure a positive birth experience, where women can make conscious choices and receive uninterrupted support throughout the labor and delivery process. Birth support during birth, use of evidence-based practices, use of non-pharmacological methods in anxiety and pain management, implementation of practices in cooperation with the woman, communication, informing the woman about the process, using positive language, and respecting privacy are the roles of health professionals in increasing birth satisfaction. The total raw score varies between 42-210. As the total score from the scale increases, the mothers' satisfaction levels with cesarean birth increase. The cut-off score 146.5.

SECONDARY OUTCOMES:
labor pain | Between 0-25th minutes of cesarean delivery
  Labor pain is a biopsychosocial process because it is a multifaceted, subjective and personal phenomenon perceived by pregnant women. The probability of experiencing pain during a cesarean section is 0.5-17% in pregnant women who undergo spinal anesthesia. Pain during a cesarean section plays an effective role in the severity of pain in the postpartum period. The severity of pain in the postpartum period has negative effects such as negative maternal bonding, postpartum depression, post-traumatic stress disorder, and prolonged hospital stay.The effectiveness of virtual reality application, a nonpharmacological method option in the management of pain perception during labor, was evaluated. Virtual reality is used as a distraction method by completely removing the individual from the area they are in. Visual analog scale was used in pain assessment. The scale in question is numbered from 0 to 10. Increasing number given to the scale indicates high pain.
blood pressure | blood pressure were measured at 3 different times: 6-12th hours before cesarean delivery, 0-25th minutes during cesarean section, and finally between 8-12th hours in the postpartum period
  A cesarean section can trigger activation of the sympathetic nervous system, leading to increased blood pressure. Blood pressure is expressed in units of pressure, also known as "mmHg" or "torr." High blood pressure is a sign of poor health.
heart rate | heart rate were measured at 3 different times: 6-12th hours before cesarean delivery, 0-25th minutes during cesarean section, and finally between 8-12th hours in the postpartum period
  A cesarean section can trigger sympathetic nervous system activation, causing an increase in heart rate. Heart rate is expressed as beats per minute (bpm). A high heart rate indicates poor health.
respiratory rate | respiratory rate were measured at 3 different times: 6-12th hours before cesarean delivery, 0-25th minutes during cesarean section, and finally between 8-12th hours in the postpartum period
  A cesarean section can trigger sympathetic nervous system activation, causing an increase in respiratory rate. Respiratory rate is expressed as the number of breaths per minute. A high respiratory rate indicates poor health.
peripheral oxygen saturation | peripheral oxygen saturation were measured at 3 different times: 6-12th hours before cesarean delivery, 0-25th minutes during cesarean section, and finally between 8-12th hours in the postpartum period
  A cesarean section can trigger sympathetic nervous system activation, leading to a decrease in peripheral oxygen saturation. Oxygen saturation is the ratio of oxygen-saturated hemoglobin to total hemoglobin in the blood and is expressed as a percentage. Approaching 100% is considered positive. Low peripheral oxygen saturation indicates poor health.
apgar scores | 1th and 5th minutes of the baby's birth
  Apgar Score Scale is a scale used to evaluate the general condition of the newborn and objectively measure the response to resuscitation practices. Apgar score is based on five clinical parameters; heart rate, respiration, muscle tone, reflex response and skin color. Each parameter is scored as 0, 1 and 2 according to predefined criteria. The minimum score that can be obtained from this scale is ''0'' and the maximum score is ''10''. An increase in the score indicates that the newborn's condition is good. Heart rate is expressed in the number of heartbeats in 1 minute and bpm. Each of these measurements will be evaluated separately. Respiration is evaluated according to whether breathing progresses regularly.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazit University, Faculty Of Health Sciences, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (4):
  • Study Protocol (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT07080281/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT07080281/SAP_001.pdf
  • Informed Consent Form: control group consent form (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT07080281/ICF_002.pdf
  • Informed Consent Form (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT07080281/ICF_003.pdf